CLINICAL TRIAL: NCT05810909
Title: Effects of Amorphous Calcium Carbonate Supplementation on Bone Health Based on Bone Mineral Density and Bone Turno-ver Markers: A Randomized, Double-Blind, Placebo-Controlled Parallel-Group Trial in Postmenopausal Women With Osteopenia
Brief Title: Effects of Amorphous Calcium Carbonate Supplementation on Bone Health in Postmenopausal Women With Osteopenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universal Integrated Corp. (Industry)
Collaborators: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: N201912029
Record Dates: First submitted 2023-03-30; First posted 2023-04-13 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Calcium; Osteopenia; Bone Mineral Density; Bone Turnover Marker
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Intervention Model Description: A Placebo-Controlled Parallel-Group Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A Randomized, Double-Blind Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACC group (Experimental): ACC group use amorphous calcium carbonate
  Interventions: Dietary Supplement: amorphous calcium carbonate/ Placebo
- control group (Placebo Comparator): control group use placebo
  Interventions: Dietary Supplement: amorphous calcium carbonate/ Placebo

INTERVENTIONS:
Dietary Supplement: amorphous calcium carbonate/ Placebo — The dosage was 1000 mg calcium carbonate (400mg calcium element) per day, and placebo (calcium carbonate change to excipient)

SUMMARY:
This research was designed in accordance to the Method for Efficacy Assessment of Health Food for Bone Heath. Changes to bone density were measured to evaluate the effectiveness of amorphous calcium carbonate in maintaining bone health.

DETAILED DESCRIPTION:
Bone comprises organic matter, predominantly protein, and inorganic matter including various mineral salts. Inappropriate nutrition profile can affect the balance of bone metabolism and cause bone loss. Of all nutrients, calcium is considered the most important for bone structure and metabolism. It is the most common deficit that affects bone health. Low dietary calcium intake can lead to negative calcium balance. Low blood calcium (< 10mg/dL) induces the release of parathyroid hormone (PTH), which activates the conversion process of 25-(OH)-D3 to physiologically active 1,25-(OH)2-D3 in kidneys. PTH and 1,25-(OH)2-D3 act jointly to change the ionic valence of hydroxyapatite, converting orthophosphate to pyrophosphate. This causes hydroxyapatite to easily dissociate and release calcium ion in order to compensate the blood calcium level. This is called bone resorption. While this physiological mechanism maintains blood calcium homeostasis, it also causes bone loss that can develop into osteoporosis. Negative calcium balance is not only caused by lack of dietary calcium, hormonal abnormality or vitamin D deficit may also lead to negative calcium balance and the development of osteoporosis. This study aims to assess the effects of UIC Amorphous Calcium on osteoporosis with "Bone Change Test" and "Calcium Bioavailability Test".

ELIGIBILITY:
Inclusion Criteria:

* Menopausal women were recruited (those who had just started menopause or less than 10 years post-menopause were preferred).

Exclusion Criteria:

* respiratory insufficiency,
* sleep apnea,
* gastroesophageal reflux,
* neurological or liver disease,
* malignant tumor, alcohol abuse,
* hysterectomy or hormonal therapy,
* and depressive symptoms.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Postmenopausal Women
Enrollment: 35 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2022-09-22 (Actual)

PRIMARY OUTCOMES:
bone density change | 6 months
  monitoring bone mineral density change and bone turnover markers change

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Wen Chien, professor, Principal Investigator — Taipei Medical University
Locations (1):
- Taipei Medical University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No